CLINICAL TRIAL: NCT01690793
Title: Measurement of Natriuretic Hormone Peptides in Exacerbation of Asthma
Acronym: acute asthma
Status: Completed | Type: Observational
Sponsor: University of South Florida (Other)
Responsible Party: Principal Investigator, Richard Lockey, prinicpal investigator, University of South Florida
Other Study IDs: acute asthma
Record Dates: First submitted 2010-08-05; First posted 2012-09-24 (Estimated); Last update posted 2015-05-28 (Estimated); Status verified 2015-05

CONDITIONS: ASTHMA
Keywords: ASTHMA; ACUTE EXACERBATION OF ASTHMA
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Biospecimen Retention: Samples With DNA — Samples of blood will be secured in the Division of Allergy/Immunology at the University of South Florida, Joy McCann Culverhouse Airways Disease Center. All samples will be appropriately coded to maintain confidentiality. Blood specimens will be held at minus 20 degrees Celsius. GENETICS SAMPLES ARE OPTIONAL
Oversight: Data Monitoring Committee: No

SUMMARY:
The investigators hypothesize that there is a statistically significant decrease of Natriuretic Hormone Peptides (NHPs) in subjects with asthma exacerbation compared to levels following treatment of an exacerbation of asthma.

DETAILED DESCRIPTION:
Overall Study Design

1. Measurement of Natriuretic Hormone Peptides in individuals suffering from exacerbation of asthma.
2. Measurement of Natriuretic Hormone Peptides 5-7 days after initiation of treatment of exacerbation of asthma.
3. Measurement of Natriuretic Hormone Peptides 10-14 days after initiation of treatment of exacerbation of asthma.

3 comparisons of Natriuretic Hormone Peptides levels will be made:

1. Exacerbation compared to 5-7 days after initiation of treatment
2. Exacerbation compared to 10-14 days after initiation of treatment
3. 5-7 days after initiation of treatment compared to 10-14 days after initiation of treatment.

Samples of blood will be secured in the Division of Allergy/Immunology at the University of South Florida, Joy McCann Culverhouse Airways Disease Center. All samples will be appropriately coded to maintain confidentiality. Blood specimens will be held at minus 20 degrees Celsius.

ELIGIBILITY:
Inclusion Criteria:

* Both genders, age 18-85.
* Females who are pregnant or lactating are not eligible.
* Read and comprehend English.
* Ability to give informed consent.
* Seen in the outpatient setting at one of the clinic.
* The subject must have a history of physician diagnosed asthma for at least 1 year and must have an exacerbation of asthma for entry into the study.

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: The Asthma Control Test score of less than 18.
  Asthma control test consists of five questions, scored 1-5 each.
Sampling Method: Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2009-02; Primary Completion 2010-12 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
The measurement of NHPs after treatment of an exacerbation of asthma | 14 days

CONTACTS AND LOCATIONS:
Locations (1):
- Usf Asthma Allergy and Immunology Cru, Tampa, Florida, United States